CLINICAL TRIAL: NCT02162368
Title: Laryngeal Mask Use in Knee-chest Position in Lumbar Surgery in Neurosurgical Patients
Status: Completed | Type: Observational
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Ricard Valero, Ricard Valero, MD, PhD, Fundacion Clinic per a la Recerca Biomédica
Other Study IDs: HCB/2014/0097
Record Dates: First submitted 2014-06-11; First posted 2014-06-12 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Airway Management; Spine Surgery; Prone Position
Keywords: laryngeal mask, prone position, spine surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Spine surgery is the most common procedure in neurosurgical setting. Some centers have chosen the patient self-position to avoid complications such as accidental extubation or loss of the iv line. The aim of our retrospective study is to describe our experience in the laryngeal mask use for airway management in patient submitted to spine surgery in neurosurgery

DETAILED DESCRIPTION:
Retrospective analysis of our experience in the last 8 years with the airway management in spine surgery in prone position. A total of 358 cases were reviewed from 2008 to 2013.

Airway management (need for LM repositioning, orotracheal intubation because of failed LM insertion), anticipated difficult airway, and airway complications were registered. Statistics were compared between groups with the t test or the χ test, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* elective spinal surgery

Exclusion Criteria:

* emergency cases
* complex spine surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent scheduled spine surgery in prone position
Sampling Method: Non-Probability Sample
Enrollment: 358 (Actual)
Dates: Start 2008-01; Primary Completion 2013-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
safety in the use of laryngeal mask in knee chest position in spine surgery | 3 years
  Analyse in a 3 years period of time, the incidence of complications in patients submitted to spinal surgery with tracheal intubation versus Laryngeal mask in prone position.

CONTACTS AND LOCATIONS:
Overall Officials: Ricard Valero, MD, PhD, Principal Investigator — Head of neuroanesthesia
Locations (1):
- Anesthesia department, Hospital Clínic de Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No